CLINICAL TRIAL: NCT00999778
Title: Optimizing Social and Communication Outcomes for Toddlers With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Connie Kasari, Professor of Psychological Studies in Education and Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1P50HD055784 (NIH)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Social and Communication Deficits in Autism; Parent and Caregiver interventions with children with Autism; Autism Spectrum Disorder; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caregiver Education Intervention (Active Comparator): 10 1:1,one hour sessions weekly for 10 weeks with parent and interventionist. Behavioral education strategies will be targeted
  Interventions: Behavioral: Caregiver-Education Intervention
- Caregiver-Mediated Intervention (Active Comparator): One hour 1:1 with parent, child and interventionist, each week, for 10 weeks social communication and joint engagement strategies will be targeted
  Interventions: Behavioral: Caregiver-Mediated Intervention

INTERVENTIONS:
Behavioral: Caregiver-Mediated Intervention — 1 (two- 1/2 jour sessions weekly) hour of intervention per week for 10 weeks in which parents and their child meet with the interventionist together using the caregiver as a means to facilitate change in their child's development
  Arms: Caregiver-Mediated Intervention
Behavioral: Caregiver-Education Intervention — The caregiver meets 1 time (1 hour each session) a week for 10 weeks with an interventionist - caregiver will receive information on child development and have the opportunity to ask questions and discuss the information vis-a-vis their own child
  Arms: Caregiver Education Intervention

SUMMARY:
This project will examine the efficacy of two different treatment approaches aimed at facilitating change in social and communications outcomes of toddlers with autism.

DETAILED DESCRIPTION:
The proposed research tests a theoretically and empirically derived treatment approach aimed at facilitating change in joint attention interactions between caregivers and their toddlers with autism. Young children with autism show impairments in engaging in joint attention skills such as pointing and showing. The importance of joint attention is underscored by data showing that these skills are important to later development of language. Yet these interaction and skills deficits have rarely been the focus of systematic intervention efforts, particularly with caregivers. Moreover, current interventions for young children wiht autism are behavioral in approach, therapist driven, and often exclude the lowest functioning and developmentally youngest children. Thus, targeting these deficits in developmentally young children using familiar caregivers may result in better language outcomes for these children.

The overarching goal of the proposed project is to rigorously test an intervention program for caregivers and their toddlers with autism that is developmentally informed, child-centered and focused on joint attention intervention with their toddlers versus mothers who receive parent education about autism and child development.

The Primary aims of this research are as follows:

* Aim 1: To determine if caregiver mediated intervention on joint engagement is superior to caregiver education on social communication and language outcomes in children.
* Aim 2: To determine if skill development in the context of caregiver child interaction transfers to interactions with classroom teachers and peers.
* Aim 3: To examine characteristics of families and children that best predict social-communication outcome.

ELIGIBILITY:
Inclusion Criteria:

* Child meets screening criteria for PDD
* Not currently enrolled in a pre-existing intervention program
* Parent is available for intervention
* Child must be ready to start in the Early Childhood Partial Hospitalization Program (ECPHP) at UCLA

Exclusion Criteria:

* Child does not have other sensory or genetic disorders
* Children already on medication on the outset, although we find few toddlers already on medication when they begin treatment. If children begin medication after treatment commences, then we will keep all informatin and data pertaining to possible medication effects and statistically convey medication use if necessary
* Co-morbidity, participant diagnosed with other diseases
* Family/participant unable to follow-up

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cognitive Assessment - Mullen Scales of Early Learning (MSEL) | Before treatment begins and at the 6 month follow up
Language Assessment - Reynell Developmental Language Scales | Before treatment begins and at 6 month follow up

SECONDARY OUTCOMES:
Language Sample - The Caregiver Child Interaction will be coded at each timepoint to obtain a 10 minute sample of the child's language transcription will yield a measure of lexical density, type-token ration and mean length of utterances | Prior to Intervention, two follow up points 3 month post intervention and 6 months post intervention
Early Social-Communication Scales; frequencies of initiating and responses of joint attention behaviors to toys and l interaction - sessions will be video taped | Before intervention, at the end of intervention and at the 3 and 6 month follow up
MacArthur Communicative Development Inventories | Before Intervention, after intervention at 3 month and 6 month follow ups
Parent Expectancy/Belief in the Intervention - assesses caregiver beliefs that the intervention is appropriate and working for the child | Before intervention and once during each phase of the intervention for total of 3 ratings (during intervention)
ADOS - The Autism Diagnostic Observation Schedule - semi-structured, standardized assessment of communication, social interaction, play and imaginative use of materials | Prior to intervention (determines eligibility) and 6 months post intervention
Generalization of skills to classroom - Observational measure to determine whether child show generalization of skill to the classroom,and in interaction with teachers & peers | Prior to intervention and once during each phase of intervention
Coding of child behaviors in classroom - using time sampling procedure, four different contexts; direct instruction, structure play, circle-time, unstructured play | during intervention
Caregiver-child interaction - A 10-minute interaction between parent and child | Pre-intervention, 3 times turing active intervention, post treatment and at 3 and 6 months follow-up
ADI-R Clinical diagnostic instrument for assessing autism in children | Prior to intervention to determine eligibility for participation in the study
Parenting Stress - The Parenting Stress Index (PSI) measuring parents reported stress associated with the care of autistic child | Prior to interventin, at the end of intervention and 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Abidin, RR, Parenting Stress Index Manual, Pediatric Psychology Press Charlottesville, VA 1983
- [Background] Adamson LB, Bakeman R, Deckner DF. The development of symbol-infused joint engagement. Child Dev. 2004 Jul-Aug;75(4):1171-87. doi: 10.1111/j.1467-8624.2004.00732.x. PMID 15260871
- [Background] Akhtar N, Dunham F, Dunham PJ. Directive interactions and early vocabulary development: the role of joint attentional focus. J Child Lang. 1991 Feb;18(1):41-9. doi: 10.1017/s0305000900013283. PMID 2010504
- [Background] Bakeman R, Adamson LB. Coordinating attention to people and objects in mother-infant and peer-infant interaction. Child Dev. 1984 Aug;55(4):1278-89. PMID 6488956
- [Background] Barnes S, Gutfreund M, Satterly D, Wells G. Characteristics of adult speech which predict children's language development. J Child Lang. 1983 Feb;10(1):65-84. doi: 10.1017/s0305000900005146. No abstract available. PMID 6841502
- [Background] Baron-Cohen S. The autistic child's theory of mind: a case of specific developmental delay. J Child Psychol Psychiatry. 1989 Mar;30(2):285-97. doi: 10.1111/j.1469-7610.1989.tb00241.x. PMID 2523408
- [Background] Curcio F. Sensorimotor functioning and communication in mute autistic children. J Autism Child Schizophr. 1978 Sep;8(3):281-92. doi: 10.1007/BF01539631. PMID 690064
- [Background] D'Amico EJ, Neilands TB, Zambarano R. Power analysis for multivariate and repeated measures designs: a flexible approach using the SPSS MANOVA procedure. Behav Res Methods Instrum Comput. 2001 Nov;33(4):479-84. doi: 10.3758/bf03195405. PMID 11816450
- [Background] Harris S, Kasari C, Sigman MD. Joint attention and language gains in children with Down syndrome. Am J Ment Retard. 1996 May;100(6):608-19. PMID 8735574
- [Background] Lovaas OI. Behavioral treatment and normal educational and intellectual functioning in young autistic children. J Consult Clin Psychol. 1987 Feb;55(1):3-9. doi: 10.1037//0022-006x.55.1.3. No abstract available. PMID 3571656
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Kasari C, Mundy P, Yirmiya N, Sigman M. Affect and attention in children with Down syndrome. Am J Ment Retard. 1990 Jul;95(1):55-67. PMID 2143659
- [Background] Kasari C, Sigman M. Linking parental perceptions to interactions in young children with autism. J Autism Dev Disord. 1997 Feb;27(1):39-57. doi: 10.1023/a:1025869105208. PMID 9018581
- [Background] Kasari C, Sigman MD, Baumgartner P, Stipek DJ. Pride and mastery in children with autism. J Child Psychol Psychiatry. 1993 Mar;34(3):353-62. doi: 10.1111/j.1469-7610.1993.tb00997.x. PMID 8463373
- [Background] Kasari C, Sigman M, Mundy P, Yirmiya N. Affective sharing in the context of joint attention interactions of normal, autistic, and mentally retarded children. J Autism Dev Disord. 1990 Mar;20(1):87-100. doi: 10.1007/BF02206859. PMID 2139025
- [Background] Kasari, C., Sigman, M., Yimiya, N., & Mundy, P., Affective Development and Communication in Children with Autism, In A.P. Kaiser & D.G. Gray (Eds) Enhancing Children's Commmunication: Research Foundations for Intervention, New York: Brookes 201-222 1993
- [Background] Arnold, SD., Elliot, M., Storoschuk, S., Pickles, A., Hellriegel, C., & Lord, C., Social Directedness and Prelinguistic Vocalization in Autism, Paper presented at the meeting of the American Academy of Child and Adolescent Psychiatry, San Antonio, TX, 1993
- [Background] Baron-Cohen, S., From Attention-Goal Psychology to Belief-Desire Psychology: The Development of a Theory of Mind and its Dysfunction, In S. Baron-Cohen, H. Hager-Flusberg & DJ Cohen (Eds), Understanding other Minds: Perspectives from Autism, Oxford, UK: Oxford University Press, 1993
- [Background] Brereton, A., & Tonge, B., Preschoolers with autism: An education and skills training programme for parents, London, UK: Jessica Kingsley Publishers, 2005
- [Background] Brown, R., A first language: the early stages, Cambridge, MA: Harvard University Press, 1973
- [Background] Bruner, J.S., From communication to language: A psychological perspective, Cognition, 3, 255-287, 1974/1975
- [Background] Bryk, A., & Raudenbush, S., Hierarchial linear models: Applications and data analysis methods, Newborn Park, CA: Sage, 1992
- [Background] Cross, T.G., Mother's speech adjustments: The contribution of selected child listener variables, in C.E. Snow and C.A. Ferguson (Eds), Talking to children: Language input and acquisition, Cambridge: Cambridge University Press, 1977
- [Background] Dawson, G., & Galpert, L., Mother's use of imitative play for facilitating social responsiveness and toy play in young autistic children, Development and Psychopathology, 2, 151-162, 1990
- [Background] Donnellan, A., & Kilman, B., Behavioral approaches to social skill development in autism: Strengths, misapplications, and alternatives, In E. Schopler & G. Mesibov (Eds), Social behavior in autism,, New York: Plenum Press, 213-215, 1986
- [Background] Harding, C.G., Setting the stage for language acquisition: Communication in the first year, In R. M. Golinkoff (Ed), The transition from prelinguistic to linguistic communication, Hillsdale, NJ: Erlbaum, 1983
- [Background] Hobson, R.P., On sharing experiences, Development and Psychopathology, 1, 197-203, 1989
- [Background] Kaiser, A., Yoder, P., & Keetz, A., Evaluating milieu teaching, In S. Warren & J Reichel (Eds) Causes and effects in communication and language intervention, Baltimore, MD: Brookes, 9-47, 1992
- [Background] Kanner, L., Autistic distrubances of affective contact, Nervous Child, 2, 273-280, 1943
- [Background] Kasari, C., Jahromi, L., Freeman, S., Paparella, T., Predictors of language growth in young children with autism. Paper presented at the Gatlinburg Conference, San Diego, CA, March 2006
- [Background] Kasari C, Paparella T, Freeman S, Jahromi LB. Language outcome in autism: randomized comparison of joint attention and play interventions. J Consult Clin Psychol. 2008 Feb;76(1):125-37. doi: 10.1037/0022-006X.76.1.125. PMID 18229990
- [Background] Kasari C, Sigman M, Mundy P, Yirmiya N. Caregiver interactions with autistic children. J Abnorm Child Psychol. 1988 Feb;16(1):45-56. doi: 10.1007/BF00910499. PMID 2966189
- [Background] Kasari, C., Sigman, M., Yirmiya, N., & Mundy, P., Affective development in children with autism, in A.P. Kaiser & D.B. Bray (Eds) Enhancing chilren's communication: Reseach foundations for intervention, New York: Brookes, 201-222, 1993
- [Background] Kasari, C., Sigman, M., & Yirmiya, N., Focused and social attention in caregiver-child interactions: A comparison of autistic, mentally retarded and nonretarded children, Development and Psychopathology, 5, 403-414, 1994
- [Background] Kellam SG, Rebok GW, Ialongo N, Mayer LS. The course and malleability of aggressive behavior from early first grade into middle school: results of a developmental epidemiologically-based preventive trial. J Child Psychol Psychiatry. 1994 Feb;35(2):259-81. doi: 10.1111/j.1469-7610.1994.tb01161.x. PMID 8188798
- [Background] Kirk, R.E., Experimental design: Procedures for the behavioral sciences (2nd ed), Pacific Grove, CA: Brooks/Cole, 1982
- [Background] Koegel RL, Firestone PB, Kramme KW, Dunlap G. Increasing spontaneous play by suppressing self-stimulation in autistic children. J Appl Behav Anal. 1974 Winter;7(4):521-8. doi: 10.1901/jaba.1974.7-521. PMID 4443320
- [Background] Koegel, R., & Koegel, L., Teaching children with autism, Baltimore: Paul H. Brookes, 1995
- [Background] Lord, C., Rutter, M.D., DiLavore, P., & Risi, S., Autism diagnostic observation schedule manual, Los Angeles, CA: Western Psychological Services, 2001
- [Background] Lord, C., Storoschuk, S., Rutter, M., & Pickles, A., Using the ADI-R to diagnose autism in preschool children with autism, Infant Mental Health Journal, 14, 234-252, 1993
- [Background] Loveland KA, Landry SH. Joint attention and language in autism and developmental language delay. J Autism Dev Disord. 1986 Sep;16(3):335-49. doi: 10.1007/BF01531663. PMID 3558291
- [Background] Fenson, L., Dale, P.S., Reznik, J.S., Thal, D., Bates, E., hartung, J.P., Pethick, S., & Reilly, J.S., The MacArthur communicative development inventories: User's guide and technical manual, San Diego, CA: Singular Publishing Group, 1993
- [Background] McEachin JJ, Smith T, Lovaas OI. Long-term outcome for children with autism who received early intensive behavioral treatment. Am J Ment Retard. 1993 Jan;97(4):359-72; discussion 373-91. PMID 8427693
- [Background] Miller JF, Chapman RS. The relation between age and mean length of utterance in morphemes. J Speech Hear Res. 1981 Jun;24(2):154-61. doi: 10.1044/jshr.2402.154. PMID 7265928
- [Background] Morales, M., Mundy, P., & Rojas, J., Following the direction of gaze and language development in 6-month olds, Infant Behavior and Development, 21, 373-377, 1998
- [Background] Mullen, E., Infant Mullen Scales of Early Learning, Cranston RI: T.O.T.A.L. Child, Inc, 1989
- [Background] Mundy, P., Gomes, A., Individual differences in joint attention skill development in the second year, Infant Behavior and Development, 21, 469-482, 1998
- [Background] Mundy, P., Kasari, C., & Sigman, M., Nonverbal communiction, affective sharing and inter-subjectivity, Infant Behavior and Development, 15, 377-381, 1992
- [Background] Mundy P, Sigman M, Kasari C. A longitudinal study of joint attention and language development in autistic children. J Autism Dev Disord. 1990 Mar;20(1):115-28. doi: 10.1007/BF02206861. PMID 2324051
- [Background] Mundy, P., Sigman, M., & Kasari, C., The theory of mind and joint-attention deficits in autism. ZIn S. Baron-Cohen, H. Tager-Flusberg, & D. Cohen (Eds), Understanding other minds: Perspectives form autism, New York: Oxford University Press, 181-203, 1993
- [Background] Mundy, P., Sigman, M., & Kasari, C., Nonverbal communication, developmental level and symptom presentation in autism, Development and Psychopathology, 6, 389-041, 1994
- [Background] Mundy P, Sigman M, Ungerer J, Sherman T. Defining the social deficits of autism: the contribution of non-verbal communication measures. J Child Psychol Psychiatry. 1986 Sep;27(5):657-69. doi: 10.1111/j.1469-7610.1986.tb00190.x. PMID 3771682
- [Background] Mundy P, Sigman M, Ungerer J, Sherman T. Nonverbal communication and play correlates of language development in autistic children. J Autism Dev Disord. 1987 Sep;17(3):349-64. doi: 10.1007/BF01487065. PMID 3654487
- [Background] Ninio, A., & Bruner, J., The achievement and antecedents of labeling, Journal of Child Language, 5, 1-15, 1978
- [Background] Nock, N.K., Kazdin, A.E., Parent expectancies for child therapy: Assessment and relation to participation in treatment, Journal of Child and Family Studies, 10, 155-189, 2001
- [Background] Odom SL, Strain PS. A comparison of peer-initiation and teacher-antecedent interventions for promoting reciprocal social interaction of autistic preschoolers. J Appl Behav Anal. 1986 Spring;19(1):59-71. doi: 10.1901/jaba.1986.19-59. PMID 3710949
- [Background] Ogletree, B.T., Communication intervention for a preverbal child with autism: A case study, Focus on Autistic Behavior, 7, 1-12, 1992
- [Background] Oke NJ, Schreibman L. Training social initiations to a high-functioning autistic child: assessment of collateral behavior change and generalization in a case study. J Autism Dev Disord. 1990 Dec;20(4):479-97. doi: 10.1007/BF02216054. PMID 2279969
- [Background] Osborne JW. Power analysis for multivariate and repeated measurements designs via SPSS: correction and extension of D'Amico, Neilands, and Zambarano (2001). Behav Res Methods. 2006 May;38(2):353-4. doi: 10.3758/bf03192787. PMID 16956112
- [Background] Paperalla, T., Pruitt, L., & Kasari, C., Joint attention in parent-autistic child dyads, Poster session at the meeting of the Society for Research in Child Development, Albuqeruqe, N, April 1999
- [Background] Ratner N, Bruner J. Games, social exchange and the acquisition of language. J Child Lang. 1978 Oct;5(3):391-401. doi: 10.1017/s0305000900002063. No abstract available. PMID 701416
- [Background] Reynell, J.K., Reynell developmental language scales (revised), Windsor, England: NFER Publishing Co, 1977
- [Background] Ricks DM, Wing L. Language, communication, and the use of symbols in normal and autistic children. J Autism Child Schizophr. 1975 Sep;5(3):191-221. doi: 10.1007/BF01538152. PMID 1174124
- [Background] Rocissano, L., & Yatchmink, Y., Joint attention in mother-toddler interaction: A study of individual variation, Marril-Palmer Quarterly, 30, 11-31, 1984
- [Background] Roeyers H, Van Oost P, Bothuyne S. Immediate imitation and joint attention in young children with autism. Dev Psychopathol. 1998 Summer;10(3):441-50. doi: 10.1017/s0954579498001680. PMID 9741676
- [Background] Rogers SJ, Lewis H. An effective day treatment model for young children with pervasive developmental disorders. J Am Acad Child Adolesc Psychiatry. 1989 Mar;28(2):207-14. doi: 10.1097/00004583-198903000-00010. PMID 2466824
- [Background] Rogosa, D., & Willett, J.B., Understanding correlates of change by modeling individual differences in growth, Psychometrika, 50, 203-228, 1985
- [Background] Rutter M. Diagnosis and definition of childhood autism. J Autism Child Schizophr. 1978 Jun;8(2):139-61. doi: 10.1007/BF01537863. No abstract available. PMID 670129
- [Background] Rutter M. Cognitive deficits in the pathogenesis of autism. J Child Psychol Psychiatry. 1983 Oct;24(4):513-31. doi: 10.1111/j.1469-7610.1983.tb00129.x. No abstract available. PMID 6630326
- [Background] Schopler E, Short A, Mesibov G. Relation of behavioral treatment to "normal functioning": comment on Lovaas. J Consult Clin Psychol. 1989 Feb;57(1):162-4. doi: 10.1037//0022-006x.57.1.162. PMID 2925968
- [Background] Schriebman, L., Austims, Newbury Park, CA: Sage, 1988
- [Background] Seibert, J., Hogan, A., & Mundy, P., Assessing interactional competencies: The Early Social-Communication Scales, Infant Mental Health Journal, 3, 244-259, 1982
- [Background] Seltzer, M., Frank, K., & Bryk, A., The metric matters: The sensitivity of conclusions concerning growth in student achievement to choice of metric, Education Evaluation and Policy Analysis, 16, 41-49, 1994
- [Background] Sigman, M., & Karsari, C., Joint attention: Its origin and role in development, Erlbaum: Hilsdale, New Jersey, 189-203, 1995
- [Background] Sigman MD, Kasari C, Kwon JH, Yirmiya N. Responses to the negative emotions of others by autistic, mentally retarded, and normal children. Child Dev. 1992 Aug;63(4):796-807. PMID 1505241
- [Background] Sigman M, Mundy P, Sherman T, Ungerer J. Social interactions of autistic, mentally retarded and normal children and their caregivers. J Child Psychol Psychiatry. 1986 Sep;27(5):647-55. doi: 10.1111/j.1469-7610.1986.tb00189.x. PMID 3771681
- [Background] Sigman, M., & Ruskin, E., Soical competence in children with autism and Down's syndrome, (in preparation)
- [Background] Sigman M, Ungerer JA. Attachment behaviors in autistic children. J Autism Dev Disord. 1984 Sep;14(3):231-44. doi: 10.1007/BF02409576. PMID 6207163
- [Background] Tomasello, M. Joint attention as social cognition, in C. Moore & P. Dunham (Eds), Joint attention: Its orgin and role in development Erlbaum: Hillsdale, New Jersey, 103-130, 1995
- [Background] Tomasello, M., The role of joimt attentional processes in early language development, Language Sciences, 10, 69-88, 1998
- [Background] Tomasello M, Farrar MJ. Joint attention and early language. Child Dev. 1986 Dec;57(6):1454-63. PMID 3802971
- [Background] Tomasello, M., Mannie, S., & Kruger, A.C., Linguistic enviornment of 1-to-2-year old twins, Developmental Psychology, 22, 169-176, 1986
- [Background] Tomasello, M., & Todd, J., Joint attention and lexical acquisition style, First Language, 4, 197-211, 1983
- [Background] Ungerer JA, Sigman M. Symbolic play and language comprehension in autistic children. J Am Acad Child Psychiatry. 1981 Spring;20(2):318-37. doi: 10.1016/s0002-7138(09)60992-4. No abstract available. PMID 6167603
- [Background] Warren SF, Kaiser AP. Incidental language teaching: a critical review. J Speech Hear Disord. 1986 Nov;51(4):291-9. doi: 10.1044/jshd.5104.291. PMID 3534460
- [Background] Wetherby AM, Prutting CA. Profiles of communicative and cognitive-social abilities in autistic children. J Speech Hear Res. 1984 Sep;27(3):364-77. doi: 10.1044/jshr.2703.364. PMID 6482406
- [Background] Whalen C, Schreibman L. Joint attention training for children with autism using behavior modification procedures. J Child Psychol Psychiatry. 2003 Mar;44(3):456-68. doi: 10.1111/1469-7610.00135. PMID 12635974
- [Background] Witte JS, Greenland S, Kim LL, Arab L. Multilevel modeling in epidemiology with GLIMMIX. Epidemiology. 2000 Nov;11(6):684-8. doi: 10.1097/00001648-200011000-00012. PMID 11055630
- [Background] Wong, C., Play and joint attention of children with autism in the preschool classroom, University of California, Los Angeles, unpublished disseratation, 2006
- [Background] Yirmiya N, Kasari C, Sigman M, Mundy P. Facial expressions of affect in autistic, mentally retarded and normal children. J Child Psychol Psychiatry. 1989 Sep;30(5):725-35. doi: 10.1111/j.1469-7610.1989.tb00785.x. PMID 2793960
- [Background] Yoder, P.J., Warren, S.F., & McCathren, R.B., Determining spoken language prognosis in children with developmental disabilities, American Journal of Speech-Language Pathology, 7, 77-87, 1998
- [Derived] Schlink A, Williams J, Pizzano M, Gulsrud A, Kasari C. Parenting stress in caregiver-mediated interventions for toddlers with autism: An application of quantile regression mixed models. Autism Res. 2022 Feb;15(2):353-365. doi: 10.1002/aur.2637. Epub 2021 Nov 19. PMID 34797038
- [Derived] Gulsrud AC, Hellemann G, Shire S, Kasari C. Isolating active ingredients in a parent-mediated social communication intervention for toddlers with autism spectrum disorder. J Child Psychol Psychiatry. 2016 May;57(5):606-13. doi: 10.1111/jcpp.12481. Epub 2015 Nov 3. PMID 26525461
- [Derived] Kasari C, Gulsrud A, Paparella T, Hellemann G, Berry K. Randomized comparative efficacy study of parent-mediated interventions for toddlers with autism. J Consult Clin Psychol. 2015 Jun;83(3):554-63. doi: 10.1037/a0039080. Epub 2015 Mar 30. PMID 25822242
- See also: UCLA Center for Autism Research and Treatment Web Site — http://www.Autism.ucla.edu